CLINICAL TRIAL: NCT02057978
Title: A Prospective Multicenter Randomized Trial to Assess the Safety and Effectiveness of EXCEL-II vs. EXCEL Sirolimus Eluting Stent for the Treatment of Patients With de Novo Coronary Artery Lesions .( CREDIT II Trial )
Brief Title: EXCEL-II Stent Vesus EXCEL Stent to Treat the Patients With de Novo Coronary Artery Lesions.
Acronym: CREDIT-II
Status: Completed | Type: Observational
Sponsor: JW Medical Systems Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CREDIT-II-131105
Record Dates: First submitted 2013-11-12; First posted 2014-02-07 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
Keywords: Late Lumen Loss; MACE; Death; TLF; Thrombosis(definite or probable )
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: None Retained — Endpoint Classification: Safety/Efficacy Study Enrollment: 416 cases [Anticipated]
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- EXCEL DES: Use EXCEL DES implatationas as control group,Implant DES for CAD cases
  Interventions: Procedure: EXCEL DES implatation
- EXCEL-II DES: EXCEL-II DES implantation as control group,Implant DES for CAD cases
  Interventions: Procedure: EXCEL-II DES implantation

INTERVENTIONS:
Procedure: EXCEL DES implatation — Implant DES for CAD cases
  Other Names: Implant DES for CAD cases
  Groups: EXCEL DES
Procedure: EXCEL-II DES implantation — Implant DES for CAD cases
  Other Names: Implant EXCEL-II DES for CAD cases
  Groups: EXCEL-II DES

SUMMARY:
The purpose of this Randomized Study to evaluate the safety and efficacy of the Excel-II DES compared to the EXCEL DES in the treatment of patients with de novo coronary artery lesions.

DETAILED DESCRIPTION:
The primary end point is to observe in-stent late lumenn loss after 9 months of the stent implantation.

This study is based on non-inferior assumption (vs. EXCEL-II V EXCEL Stent), requring all of end points reach statictic significance.

Quality assurance plan that addresses data validation and registry procedures, including any plans for site monitoring and auditing.

Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (e.g., medical records, paper or electronic case report forms, or interactive voice response systems).

Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information if used and normal ranges if relevant.

Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect.

Plan for missing data to address situations where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan.

ELIGIBILITY:
Inclusion criteria:

1.18yrs≤Age≤75yrs . 2.stability and unstable angina pectoris (AP), chronic myocardial infarction (OMI) or confirmed myocardial ischemia; 3.De novo lesion at native coronary artery(Up to two target lesions). 4.Lesion length ≤32mm. 5.RVD 2.5mm～4.0mm. 6.DS%≥70% by visual test. 7.Coronary artery bypass surgery (coronary artery bypass grafting) patients. 8.Subjects are willing to follow the specified requirements follow-up. 9.To understand the purpose of the trial and willing to sign informed consent and accept clinical follow-up.

Exclusion Criteria:

1. AMI within 7 days.
2. CTO (TIMI 0), the left main lesion, ostial lesion and transplant vascular lesions, the bifurcation lesion (reference collateral blood vessel diameter of 2.5 mm or higher), stent restenosis lesions and to deal with three pathological changes;
3. Severe calcified lesion unable to predilate.
4. The distortion of the stent was hampered by lesions.
5. NYHA≥Ⅲ or LVEF<40%.
6. Prior PCI within 1 year.
7. Pregnancy or lactation, and planning pregnancy or lactation.
8. Subjects have bleeding tendency or blood coagulation dysfunction or PCI contraindications, or anticoagulant therapy taboo or can't continue to take DAPT at least 1 year.
9. There are other diseases (such as cancer,malignant tumor ,congestive heart failure,organ transplantation or candidate) or abuse history (alcohol cocaine heroin, etc.), scheme compliance is poor, interference related data explanation or the limited life (< 1 year).
10. To aspirin heparin clopidogrel cobalt chromium alloy rapamycin PLA polymer contrast agent of one of allergy.
11. Serious liver and kidney function are not complete subject(ALT and AST were three times greater than the upper limit of normal).
12. Before enrolling to participate in other clinical trials and not reached the primary endpoint.
13. Non-compliant subject and could not finish the trial in accordance with the requirements of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will plan for a total of 416 patients with primary, in situ coronary artery lesions (all of the patients was selected in different blood vessels, a total of up to two target disease Variable and each target lesion 1 stents, such as placing stents need more than one in the operation, require the use of the same brand of stents, mix does not recommend the same patients Other brand support, unless save extra stents.) Choose lesions reference diameter of 2.5 mm to 2.5 mm (visual), each lesion length 32 mm or less (visual), participants must conform to the standard can be selected.
Sampling Method: Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2013-12-08 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
9 months in-stent late lumen loss | 9 months
  To observe in-stent late lumen loss after 9 months of stent implantation

SECONDARY OUTCOMES:
9-m in-segment diameter restenosis rate | 9 months
  9-m in stent, proximal stent edge, the distal edge segment defined in the restenosis rate, 9-m after lesions within the segment late lumen loss percentage and the diameter of the restenosis degree
Device success rates , lesion success rates , clinical success rates Device, lesion, & clinical success rates Device, lesion, & clinical success rates Target Lesion Failure | 1m,6m,9m,12m,18m and annually to 5years
  Device oriented composite of cardiac death, MI, or ischemia-driven TLR at 1m, 6m, 12m,18m and annually up to 5 yrs
Rate of stent thrombosis | 1m,6m,9m,12m,18m and annually up to 5 yrs
  Definite and probable stent thrombosis according to ARC defination

CONTACTS AND LOCATIONS:
Overall Officials: Han Yaling, PhD, Principal Investigator — Shenyang Northern Hospital
Locations (1):
- Shenyang Northern Hospital, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Xu K, Han Y, Xu B, Yang Y, Wang G, Li H, Sun Y, Tao L, Wang H, Yuan Z, Liu H, Liu J, Jia Y, Ma G, Fu G, Li X, Li S, Wang S, Pu K; CREDIT 2 Investigators. Efficacy and safety of a second-generation biodegradable polymer sirolimus-eluting stent: One-year results of the CREDIT 2 trial. Cardiovasc Ther. 2018 Jun;36(3):e12327. doi: 10.1111/1755-5922.12327. Epub 2018 Mar 25. PMID 29493880